CLINICAL TRIAL: NCT05245539
Title: A Randomized, Double-Blind Trial to Study the Effect of CVL-231 on 24-Hour Ambulatory Blood Pressure in Participants With Schizophrenia
Brief Title: Trial to Study the Effect of CVL-231 on 24-Hour Ambulatory Blood Pressure in Participants With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVL-231-1005
Record Dates: First submitted 2022-01-27; First posted 2022-02-18 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Blood Pressure; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CVL-231 Dose Level 1 (Experimental): 10 mg once daily
  Interventions: Drug: CVL-231
- CVL-231 Dose Level 2 (Experimental): 30 mg once daily
  Interventions: Drug: CVL-231

INTERVENTIONS:
Drug: CVL-231 — CVL-231 is a brain penetrant mAChR activator that selectively binds to the M4 mAChR subtype while sparing other muscarinic receptor subtypes (M1, M2, M3, and M5). CVL-231 is being developed for treatment of psychosis in schizophrenia.

SUMMARY:
The purpose of this trial is to characterize the effects of 2 oral doses (over 8 weeks total) of CVL-231 on ambulatory blood pressure and heart rate in patients with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, ages 30 to 60 years, inclusive, at the time of signing the ICF.
* Primary diagnosis of schizophrenia per DSM-5, as confirmed by the MINI version 7.0.2.
* PANSS Total Score ≤70 at the time of signing the ICF and Check-in (Day -5).

Exclusion Criteria:

* Current DSM-5 diagnosis other than schizophrenia including, but not limited to, mental retardation; schizoaffective disorder; major depressive disorder; schizophreniform disorder; psychotic depression; bipolar disorder; post-traumatic stress disorder; generalized anxiety disorder, obsessive compulsive disorder, eating disorders (bulimia, anorexia), or other anxiety disorders as a primary diagnosis (Note: Anxiety symptoms secondary to schizophrenia are allowed); delirium, dementia, amnestic, or other cognitive disorders. Acute depressive symptoms within 30 days prior to signing the ICF that require treatment with an antidepressant are exclusory. Additional excluded conditions include borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Any of the following:

  * Schizophrenia considered resistant/refractory (defined as failure to respond to 2 or more courses of adequate pharmacological treatment) to antipsychotic treatment by history
  * History of failure to respond to clozapine
  * Response to clozapine treatment only
* History of extrapyramidal symptoms treated with a medication that required dose modification and/or new treatment within 6 months prior to signing the ICF.
* Current or past history of significant cardiovascular disease including any of the following: ischemic heart disease, myocardial infarction, cardiac valvulopathy, cardiac surgery revascularization (coronary artery bypass grafting) or stenting or percutaneous transluminal coronary angioplasty), hypertension, receiving medications to treat hypertension, orthostatic hypotension, angina, unstable angina, cerebrovascular accident or stroke or transient ischemic attack, pacemaker, atrial fibrillation, atrial flutter, paroxysmal atrial tachycardia, or non-sustained or sustained ventricular tachycardia, pulmonary arterial hypertension, sick sinus syndrome, Type 2 second-degree or third-degree atrioventricular block, congestive heart failure, personal or family history of sudden death or long QT syndrome, unexplained syncope or syncope within the last 3 years regardless of etiology.
* 12-lead ECG demonstrating any of the following at the Screening Visit or at Check-in (Day -5):

  * QTcF interval >450 ms
  * QRS interval >120 ms (unless right bundle branch block)
  * PR interval >200 ms
  * LVH with ST depressions and/or T wave inversions in leads with relatively tall R waves (ie, LVH with associated ST-T wave abnormalities)
  * Type 2 second-degree or third-degree atrioventricular block
  * Heart rate <45 bpm or >90 bpm
  * Abnormal acute ECG changes (such as clinically significant ST depression or elevation or T wave inversion)
  * Abnormal heart rhythm (atrial fibrillation and atrial flutter)
* Blood pressure measurements demonstrating any of the following at the Screening Visit and at Check-in (Day -5):

  * Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg

    o Blood pressure will be measured in a seated position after at least 3 minutes of rest. The average of 3 measurements will be used to determine eligibility.
  * Orthostatic hypotension, defined as a decrease of ≥20 mmHg in systolic blood pressure after at least 2 minutes of standing compared with the average of the resting supine blood pressure measurement

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline to Week 8 in the 24-hour ambulatory SBP (Systolic Blood Pressure) | Baseline to week 8

SECONDARY OUTCOMES:
Mean changes from Baseline to Weeks 4 and 8 in ambulatory SBP during daytime period | At weeks 4 and 8
Mean changes from Baseline to Weeks 4 and 8 in ambulatory SBP during nighttime period | At weeks 4 and 8
Mean change from Baseline to Week 4 in the 24-hour ambulatory SBP | At week 4
Mean change from Baseline to Weeks 4 and 8 in the 24-hour ambulatory DBP (Diastolic blood pressure) | At week 8
Mean change from Baseline to Weeks 4 and 8 in the 24-hour ambulatory HR (Heart rate) | At weeks 4 and 8
Number of treatment-emergent adverse events | Screening through day 84
Frequency of clinically significant changes in electrocardiograms | Baseline through day 84
Frequency of clinically significant changes in clinical laboratory assessments | Baseline through day 84
Frequency of clinically significant changes in vital sign measurements | Baseline through day 84
Frequency of clinically significant changes in physical examination results | Baseline through day 84
Frequency of clinically significant changes in neurological examination results | Baseline through day 84
Frequency of clinically significant findings in suicidality assessed using the C-SSRS (Columbia Suicide Severity Rating Scale) | Baseline through day 84
Frequency of clinically significant findings in extrapyramidal symptoms evaluated using the SAS (Simpson Angus Scale) | Baseline through day 84
Frequency of clinically significant findings in extrapyramidal symptoms evaluated using the AIMS (Abnormal Involuntary Movement Scale) | Baseline through day 84
Frequency of clinically significant findings in extrapyramidal symptoms evaluated using the BARS (Barnes Akathisia Rating Scale) | Baseline through day 84
Steady state CVL-231 Peak Plasma Concentration (Cmax) for CVL-231 and Metabolite (PF-06892787) | Baseline through day 84
Area under the plasma concentration-time curve over dosing interval (AUCτ) for CVL-231 and Metabolite (PF-06892787) | Baseline through day 84

CONTACTS AND LOCATIONS:
Overall Officials: Erica Koenig, PhD, Study Director — Cerevel Therapeutics, LLC
Locations (10):
- United States (10):
  - Pillar Clinical Research LLC, Bentonville, Arkansas
  - Woodland International Research Group LLC - ERG - PPDS, Little Rock, Arkansas
  - Collaborative NeuroScience Research, LLC - Torrance - Apex - PPDS, Long Beach, California
  - Innovative Clinical Research, Inc - ClinEdge - PPDS, Miami, Florida
  - Uptown Research Institute LLC, Chicago, Illinois
  - Pillar Clinical Research LLC, Lincolnwood, Illinois
  - Hassman Research Institute - Apex - PPDS, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Community Clinical Research, Austin, Texas
  - Pillar Clinical Research LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No